CLINICAL TRIAL: NCT04881357
Title: Evaluation of Antiplaque and Antigingivitis Effects of the New "Lacer Oros Acción Integral" Mouth Rinse Formulation.
Brief Title: Antiplaque/Antigingivitis Effect of Lacer Oros Integral
Acronym: LacerINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Lacer S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20/750-EC_X
Record Dates: First submitted 2021-04-26; First posted 2021-05-11 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Periodontitis; Dental Plaque; Gingival Inflammation
MeSH Terms: conditions — Periodontitis; Dental Plaque; Gingivitis | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: pilot, parallel, double-blind, randomized, placebo-controlled, 12-week, clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will use three times daily a provided manual toothbrush with a sodium fluoride dentifrice, followed by the use of the test mouth rinse (Lacer Oros Acción Integral - new formula, Barcelona, Spain).
  Interventions: Other: test mouth rinse (Lacer Oros Acción Integral - new formula, Barcelona, Spain).
- Control Group (Placebo Comparator): The control group will use three times daily a provided manual toothbrush with a sodium fluoride dentifrice, followed by the use of the control mouth rinse (Lacer Oros Acción Integral - new formula, without active ingredients, Barcelona, Spain).
  Interventions: Other: control group

INTERVENTIONS:
Other: test mouth rinse (Lacer Oros Acción Integral - new formula, Barcelona, Spain). — The experimental group will use three times daily a provided manual toothbrush with a sodium fluoride dentifrice, followed by the use of the test mouth rinse (Lacer Oros Acción Integral - new formula, Barcelona, Spain).
  Arms: Experimental Group
Other: control group — The control group will use three times daily a provided manual toothbrush with a sodium fluoride dentifrice, followed by the use of the control mouth rinse (Lacer Oros Acción Integral - new formula, without active ingredients, Barcelona, Spain).
  Arms: Control Group

SUMMARY:
Background; A new mouth rinse formulation ("Lacer Oros Acción Integral", Lacer SA, Barcelona, Spain) has been recently proposed, including O-Cymen-5-ol, potassium nitrate, zinc chloride, dipotassium glycyrrhizate, sodium fluoride, panthenol and xylitol, within its ingredients. Thus, it may be relevant to test the efficacy of this new "Lacer Oros Acción Integral" mouth rinse formulation in a RCT.

Primary Objective: The primary objective of this RCT will be to evaluate the antiplaque/antigingivitis effects of the test mouth rinse.

Population: Consecutive subjects in supportive periodontal therapy (SPT) will be screened at the Post-Graduate Periodontal Clinic in the University Complutense, Madrid, and enrolled in the clinical trial if they are periodontitis patients, already enrolled in a SPT, for at least 6 months, systemically healthy, with moderate gingival inflammation and complains of dentin hypersensitivity.

Study design: pilot, parallel, double-blind, randomized, placebo-controlled, 12-week, clinical trial

Intervention: The experimental group will use three times daily a provided manual toothbrush with a sodium fluoride dentifrice, followed by the use of the test mouth rinse (Lacer Oros Acción Integral - new formula, Barcelona, Spain). The control group will use three times daily a provided manual toothbrush with a sodium fluoride dentifrice, followed by the use of the control mouth rinse (Lacer Oros Acción Integral - new formula, without active ingredients, Barcelona, Spain).

Visits: Screening, baseline, 2 and 12 weeks.

Outcomes: Periodontal clinical outcomes (plaque levels, gingival condition, probing pocket depth), Stainign, Microbiological outcomes (culture and qPCR). Patient reported outcomes, compliance, adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* 35-64 years old.
* Periodontitis patients, already enrolled in a SPT, for at least 6 months, and the last SPT visit in the previous 6 months.
* Systemically healthy, following the criteria of the American Society of Anesthesiologists (ASA), for patients ASA type I or II (see also exclusion criteria).
* Presence of at least three evaluable teeth in each quadrant.
* Moderate gingival inflammation (≥40% bleeding on marginal probing, BOMP) (Van der Weijden, Timmerman, Nijboer, Reijerse, & Van der Velden, 1994) and Turesky plaque index ≥1.5. Also 2017 World Workshop criteria and bleeding on probing (BOP) (Ainamo & Bay, 1975) criteria will be considered. The primary criteria will be BOP ≥30% and Turesky plaque index ≥1.5
* No orthodontic banding or removable prosthesis.
* Subjects willing to participate and comply with the requirements of the study.
* Complains of dentin hypersensitivity in, at least, one evaluable tooth. Dentin hypersensitivity will be confirmed with evaporative sensitivity (Schiff et al., 1994), with a minimum score of 2-3 (West et al., 2013), although a score of 1 will also be considered as adequate. In order to be eligible, the selected tooth must not have a current desensitizing therapy, must not have been restored in the last 3 moths, or have a crown or a big restoration. Only incisors, canines and premolars will be considered (Holland, Narhi, Addy, Gangarosa, & Orchardson, 1997).

Exclusion Criteria:

* Untreated or uncontrolled periodontitis
* Regular use of antiseptic-containing and/or anti-hypersensitivity mouth rinses.
* Antibiotic intake within the previous month.
* Excessive exposure to acids (eating disorders, chronic regurgitation).
* Chronic use of analgesic or anti-inflammatory drugs.
* Pregnant women.
* Any adverse medical history (diabetes, osteoporosis, immunosuppression…) or long-term medication (chemotherapy and immunosuppression treatment; pharmacological treatment associated with gingival overgrowth such as the use of phenytoin, phenobarbital, lamotrigine, vigabatrin, ethosuximide, topiramate, primidone, nifedipine, amlodipine, verapamil, cyclosporine) influencing gingival conditions.
* Conditions which requires antibiotic prophylaxis (infectious endocarditis, cardiac valve prosthesis…).

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-04 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Change in BOP (Baseline-12 weeks) | Change from baseline to 12 weeks
  Gingival Bleeding Index (Ainamo & Bay, 1975), by dichotomously assessing bleeding after gentle probing.

SECONDARY OUTCOMES:
Change in BOP (Baseline-6 weeks) | Change from baseline to 6 weeks
  Gingival Bleeding Index (Ainamo & Bay, 1975), by dichotomously assessing bleeding after gentle probing.
Change in BOP (6-12 weeks) | Change from 6 to 12 weeks
  Gingival Bleeding Index (Ainamo & Bay, 1975), by dichotomously assessing bleeding after gentle probing.
BOP_baseline | Baseline
  Gingival Bleeding Index (Ainamo & Bay, 1975), by dichotomously assessing bleeding after gentle probing.
BOP_6 weeks | 6 weeks
  Gingival Bleeding Index (Ainamo & Bay, 1975), by dichotomously assessing bleeding after gentle probing.
BOP_12 weeks | 12 weeks
  Gingival Bleeding Index (Ainamo & Bay, 1975), by dichotomously assessing bleeding after gentle probing.
BOMP_baseline | Baseline
  The BOMP index by recording the presence or absence of bleeding within 30 seconds of probing on a scale 0-2 (Lie, Timmerman, Van der Velden, & Van der Weijden, 1998; Van der Weijden, Timmerman, Nijboer, et al., 1994).
BOMP_6 weeks | 6 weeks
  The BOMP index by recording the presence or absence of bleeding within 30 seconds of probing on a scale 0-2 (Lie, Timmerman, Van der Velden, & Van der Weijden, 1998; Van der Weijden, Timmerman, Nijboer, et al., 1994).
BOMP_12 weeks | 12 weeks
  The BOMP index by recording the presence or absence of bleeding within 30 seconds of probing on a scale 0-2 (Lie, Timmerman, Van der Velden, & Van der Weijden, 1998; Van der Weijden, Timmerman, Nijboer, et al., 1994).
Change in BOMP (Baseline-12 weeks) | Change from baseline to 12 weeks
  The BOMP index by recording the presence or absence of bleeding within 30 seconds of probing on a scale 0-2 (Lie, Timmerman, Van der Velden, & Van der Weijden, 1998; Van der Weijden, Timmerman, Nijboer, et al., 1994).
Change in BOMP (Baseline-6 weeks) | Change from baseline to 6 weeks
  The BOMP index by recording the presence or absence of bleeding within 30 seconds of probing on a scale 0-2 (Lie, Timmerman, Van der Velden, & Van der Weijden, 1998; Van der Weijden, Timmerman, Nijboer, et al., 1994).
Change in BOMP (6-12 weeks) | Change from 6 to 12 weeks
  The BOMP index by recording the presence or absence of bleeding within 30 seconds of probing on a scale 0-2 (Lie, Timmerman, Van der Velden, & Van der Weijden, 1998; Van der Weijden, Timmerman, Nijboer, et al., 1994).
Change in Dental Plaque (Baseline-12 weeks) | Change from baseline to 12 weeks
  Dental plaque will be assessed using a disclosing solution (PlacControl®, Dentaid, Barcelona, Spain) with the Turesky et al. (Turesky, Gilmore, & Glickman, 1970) modification of the Quigley and Hein index (Quigley & Hein, 1962), scored at six sites per tooth.
Change in Dental Plaque (Baseline-6 weeks) | Change from baseline to 6 weeks
  Dental plaque will be assessed using a disclosing solution (PlacControl®, Dentaid, Barcelona, Spain) with the Turesky et al. (Turesky, Gilmore, & Glickman, 1970) modification of the Quigley and Hein index (Quigley & Hein, 1962), scored at six sites per tooth.
Change in Dental Plaque (6-12 weeks) | Change from 6 to 12 weeks
  Dental plaque will be assessed using a disclosing solution (PlacControl®, Dentaid, Barcelona, Spain) with the Turesky et al. (Turesky, Gilmore, & Glickman, 1970) modification of the Quigley and Hein index (Quigley & Hein, 1962), scored at six sites per tooth.
Dental Plaque_Baseline | Baseline
  Dental plaque will be assessed using a disclosing solution (PlacControl®, Dentaid, Barcelona, Spain) with the Turesky et al. (Turesky, Gilmore, & Glickman, 1970) modification of the Quigley and Hein index (Quigley & Hein, 1962), scored at six sites per tooth.
Dental Plaque_6 weeks | 6 weeks
  Dental plaque will be assessed using a disclosing solution (PlacControl®, Dentaid, Barcelona, Spain) with the Turesky et al. (Turesky, Gilmore, & Glickman, 1970) modification of the Quigley and Hein index (Quigley & Hein, 1962), scored at six sites per tooth.
Dental Plaque_12 weeks | 12 weeks
  Dental plaque will be assessed using a disclosing solution (PlacControl®, Dentaid, Barcelona, Spain) with the Turesky et al. (Turesky, Gilmore, & Glickman, 1970) modification of the Quigley and Hein index (Quigley & Hein, 1962), scored at six sites per tooth.
Staining of teeth_baseline | Baseline
  Staining of teeth will be scored using the Gründemann modification of the stain index (GMSI) (Gründemann, Timmerman, IJzerman, Van der Weijden, & Van der Weijden, 2000), recorded at nine areas per tooth (three mesial, three medial, three distal) (Koertge, Gunsolley, Domke, & Nelson, 1993). Stain will be graded using the intensity stain index of Lobene (Lobene, 1968). Presence of staining will be assessed in the upper and lower anterior buccal sites, by evaluating standardized clinical photographs by two calibrated examiners.
Staining of teeth_6 weeks | 6 weeks
  Staining of teeth will be scored using the Gründemann modification of the stain index (GMSI) (Gründemann, Timmerman, IJzerman, Van der Weijden, & Van der Weijden, 2000), recorded at nine areas per tooth (three mesial, three medial, three distal) (Koertge, Gunsolley, Domke, & Nelson, 1993). Stain will be graded using the intensity stain index of Lobene (Lobene, 1968). Presence of staining will be assessed in the upper and lower anterior buccal sites, by evaluating standardized clinical photographs by two calibrated examiners.
Staining of teeth_12 weeks | 12 weeks
  Staining of teeth will be scored using the Gründemann modification of the stain index (GMSI) (Gründemann, Timmerman, IJzerman, Van der Weijden, & Van der Weijden, 2000), recorded at nine areas per tooth (three mesial, three medial, three distal) (Koertge, Gunsolley, Domke, & Nelson, 1993). Stain will be graded using the intensity stain index of Lobene (Lobene, 1968). Presence of staining will be assessed in the upper and lower anterior buccal sites, by evaluating standardized clinical photographs by two calibrated examiners.
Probing pocket depth_baseline | Baseline
  At six sites per tooth, with a millimetre periodontal probe (North Carolina)
Probing pocket depth_6 weeks | 6 weeks
  At six sites per tooth, with a millimetre periodontal probe (North Carolina)
Probing pocket depth_12 weeks | 12 weeks
  At six sites per tooth, with a millimetre periodontal probe (North Carolina)
Recession_baseline | Baseline
  At six sites per tooth, with a millimetre periodontal probe (North Carolina)
Recession_6 weeks | 6 weeks
  At six sites per tooth, with a millimetre periodontal probe (North Carolina)
Recession_12 weeks | 12 weeks
  At six sites per tooth, with a millimetre periodontal probe (North Carolina)
Dentin hypersensitivity_baseline | Baseline
  Dentin hypersensitivity will be explored by means of evaporative stimulus, with two distinct assessments: an objective assessment, using the Schiff scale (Schiff et al., 1994): a subjective assessment, using the Visual Analogue Scales (VAS), as reported by the patient. Dentin hypersensitivity will be scored in just one tooth, identified according to selection criteria, listed in the inclusion criteria. The same tooth will be also scored in the follow up visits. If the patient identifies more than one tooth with dentin hypersensitivity at baseline, the one with a higher level of pain (according to the patient evaluation), will be selected. The clinician will take the final decision concerning the selected tooth.
Dentin hypersensitivity_6 weeks | 6 weeks
  Dentin hypersensitivity will be explored by means of evaporative stimulus, with two distinct assessments: an objective assessment, using the Schiff scale (Schiff et al., 1994): a subjective assessment, using the Visual Analogue Scales (VAS), as reported by the patient. Dentin hypersensitivity will be scored in just one tooth, identified according to selection criteria, listed in the inclusion criteria. The same tooth will be also scored in the follow up visits. If the patient identifies more than one tooth with dentin hypersensitivity at baseline, the one with a higher level of pain (according to the patient evaluation), will be selected. The clinician will take the final decision concerning the selected tooth.
Dentin hypersensitivity_12 weeks | 12 weeks
  Dentin hypersensitivity will be explored by means of evaporative stimulus, with two distinct assessments: an objective assessment, using the Schiff scale (Schiff et al., 1994): a subjective assessment, using the Visual Analogue Scales (VAS), as reported by the patient. Dentin hypersensitivity will be scored in just one tooth, identified according to selection criteria, listed in the inclusion criteria. The same tooth will be also scored in the follow up visits. If the patient identifies more than one tooth with dentin hypersensitivity at baseline, the one with a higher level of pain (according to the patient evaluation), will be selected. The clinician will take the final decision concerning the selected tooth.
Patient reported outcomes-1_6 weeks | 6 weeks
  A predefined questionnaire will be filled by the patient, on product usage and perceptions, including nine different questions.
  Question 1: Mouth rinse flavor (1: very bad; 10: very good).
Patient reported outcomes-1_12 weeks | 12 weeks
  A predefined questionnaire will be filled by the patient, on product usage and perceptions, including nine different questions.
  Question 1: Mouth rinse flavor (1: very bad; 10: very good).
Patient reported outcomes-2_6 weeks | 6 weeks
  A predefined questionnaire will be filled by the patient, on product usage and perceptions, including nine different questions.
  Question 2: How much time does the mouth rinse flavor lasts in your mouth (1: very low; 10: too much)
Patient reported outcomes-2_12 weeks | 12 weeks
  A predefined questionnaire will be filled by the patient, on product usage and perceptions, including nine different questions.
  Question 2: How much time does the mouth rinse flavor lasts in your mouth (1: very low; 10: too much)
Patient reported outcomes-3_6 weeks | 6 weeks
  A predefined questionnaire will be filled by the patient, on product usage and perceptions, including nine different questions.
  Question 3: Which is your perception of the food and drinks flavor when using the mouth rinse (1: much worse, 10: better).
Patient reported outcomes-3_12 weeks | 12 weeks
  A predefined questionnaire will be filled by the patient, on product usage and perceptions, including nine different questions.
  Question 3: Which is your perception of the food and drinks flavor when using the mouth rinse (1: much worse, 10: better).
Patient reported outcomes-4_6 weeks | 6 weeks
  A predefined questionnaire will be filled by the patient, on product usage and perceptions, including nine different questions.
  Question 4: Do you notice the teeth and the mucosa more sensitive after using the mouth rinse (1: no, absolutely; 10: yes, much more).
Patient reported outcomes-4_12 weeks | 12 weeks
  A predefined questionnaire will be filled by the patient, on product usage and perceptions, including nine different questions.
  Question 4: Do you notice the teeth and the mucosa more sensitive after using the mouth rinse (1: no, absolutely; 10: yes, much more).
Patient reported outcomes-5_6 weeks | 6 weeks
  A predefined questionnaire will be filled by the patient, on product usage and perceptions, including nine different questions.
  Question 5: Do you notice a drier mouth after using the mouth rinse (1: no, absolutely; 10: yes, much more).
Patient reported outcomes-5_12 weeks | 12 weeks
  A predefined questionnaire will be filled by the patient, on product usage and perceptions, including nine different questions.
  Question 5: Do you notice a drier mouth after using the mouth rinse (1: no, absolutely; 10: yes, much more).
Patient reported outcomes-6_6 weeks | 6 weeks
  A predefined questionnaire will be filled by the patient, on product usage and perceptions, including nine different questions.
  Question 6: Do you notice burning feeling after using the mouth rinse (1: no, absolutely; 10: yes, much more).
Patient reported outcomes-6_12 weeks | 12 weeks
  A predefined questionnaire will be filled by the patient, on product usage and perceptions, including nine different questions.
  Question 6: Do you notice burning feeling after using the mouth rinse (1: no, absolutely; 10: yes, much more).
Patient reported outcomes-7_6 weeks | 6 weeks
  A predefined questionnaire will be filled by the patient, on product usage and perceptions, including nine different questions.
  Question 7: Do you notice some staining on the teeth or tongue due to the use of the mouth rinse (1: no, absolutely; 10: yes, much more).
Patient reported outcomes-7_12 weeks | 12 weeks
  A predefined questionnaire will be filled by the patient, on product usage and perceptions, including nine different questions.
  Question 7: Do you notice some staining on the teeth or tongue due to the use of the mouth rinse (1: no, absolutely; 10: yes, much more).
Patient reported outcomes-8_6 weeks | 6weeks
  A predefined questionnaire will be filled by the patient, on product usage and perceptions, including nine different questions.
  Question 8: Which is your general opinion after using the mouth rinse in this study (1: very bad; 10: very good).
Patient reported outcomes-8_12 weeks | 12 weeks
  A predefined questionnaire will be filled by the patient, on product usage and perceptions, including nine different questions.
  Question 8: Which is your general opinion after using the mouth rinse in this study (1: very bad; 10: very good).
Patient reported outcomes-9_6 weeks | 6 weeks
  A predefined questionnaire will be filled by the patient, on product usage and perceptions, including nine different questions.
  Question 9: Do you think that the mouth rinse use has improved your mouth health (1: no absolutely; 10: yes, much more).
Patient reported outcomes-9_12 weeks | 12 weeks
  A predefined questionnaire will be filled by the patient, on product usage and perceptions, including nine different questions.
  Question 9: Do you think that the mouth rinse use has improved your mouth health (1: no absolutely; 10: yes, much more).
Compliance_6 weeks | 12 weeks
  The study coordinator will collect, at each study visit, the compliance forms, filled by the patients, as well as the empty and unused mouth rinse bottles.
Compliance_12 weeks | 12 weeks
  The study coordinator will collect, at each study visit, the compliance forms, filled by the patients, as well as the empty and unused mouth rinse bottles.
Total counts (CFU/ml)_Baseline | Baseline
  Four sites will be selected, one per quadrant, based on presence of bleeding during the screening visit. The same sites will be sampled at the follow-up visit. These sites will be isolated with cotton rolls and dried gently with sprayed air. Two consecutive sterile paper points (medium size, Maillefer, Ballaigues, Switzerland) will be inserted as deep as possible into the sulcus, and leave in place for 10 seconds. The paper points will be transferred to a vial containing 1.5 mL of reduced transport fluid (Syed & Loesche, 1972), and pooled with the other paper points.
  The vial will be sent to the laboratory and processed for culture and qPCR
Total counts (CFU/ml)_6 weeks | 6 weeks
  Four sites will be selected, one per quadrant, based on presence of bleeding during the screening visit. The same sites will be sampled at the follow-up visit. These sites will be isolated with cotton rolls and dried gently with sprayed air. Two consecutive sterile paper points (medium size, Maillefer, Ballaigues, Switzerland) will be inserted as deep as possible into the sulcus, and leave in place for 10 seconds. The paper points will be transferred to a vial containing 1.5 mL of reduced transport fluid (Syed & Loesche, 1972), and pooled with the other paper points.
  The vial will be sent to the laboratory and processed for culture and qPCR
Total counts (CFU/ml)_12 weeks | 12 weeks
  Four sites will be selected, one per quadrant, based on presence of bleeding during the screening visit. The same sites will be sampled at the follow-up visit. These sites will be isolated with cotton rolls and dried gently with sprayed air. Two consecutive sterile paper points (medium size, Maillefer, Ballaigues, Switzerland) will be inserted as deep as possible into the sulcus, and leave in place for 10 seconds. The paper points will be transferred to a vial containing 1.5 mL of reduced transport fluid (Syed & Loesche, 1972), and pooled with the other paper points.
  The vial will be sent to the laboratory and processed for culture and qPCR
Proportion of periodontal pathogens (%)_Baseline | Baseline
  Four sites will be selected, one per quadrant, based on presence of bleeding during the screening visit. The same sites will be sampled at the follow-up visit. These sites will be isolated with cotton rolls and dried gently with sprayed air. Two consecutive sterile paper points (medium size, Maillefer, Ballaigues, Switzerland) will be inserted as deep as possible into the sulcus, and leave in place for 10 seconds. The paper points will be transferred to a vial containing 1.5 mL of reduced transport fluid (Syed & Loesche, 1972), and pooled with the other paper points.
  The vial will be sent to the laboratory and processed for culture and qPCR. Proportions of microbiota would be calculated as counts of the pathogen/total counts.
Proportion of periodontal pathogens (%)_6 weeks | 6 weeks
  Four sites will be selected, one per quadrant, based on presence of bleeding during the screening visit. The same sites will be sampled at the follow-up visit. These sites will be isolated with cotton rolls and dried gently with sprayed air. Two consecutive sterile paper points (medium size, Maillefer, Ballaigues, Switzerland) will be inserted as deep as possible into the sulcus, and leave in place for 10 seconds. The paper points will be transferred to a vial containing 1.5 mL of reduced transport fluid (Syed & Loesche, 1972), and pooled with the other paper points.
  The vial will be sent to the laboratory and processed for culture and qPCR. Proportions of microbiota would be calculated as counts of the pathogen/total counts.
Proportion of periodontal pathogens (%)_12 weeks | 12 weeks
  Four sites will be selected, one per quadrant, based on presence of bleeding during the screening visit. The same sites will be sampled at the follow-up visit. These sites will be isolated with cotton rolls and dried gently with sprayed air. Two consecutive sterile paper points (medium size, Maillefer, Ballaigues, Switzerland) will be inserted as deep as possible into the sulcus, and leave in place for 10 seconds. The paper points will be transferred to a vial containing 1.5 mL of reduced transport fluid (Syed & Loesche, 1972), and pooled with the other paper points.
  The vial will be sent to the laboratory and processed for culture and qPCR. Proportions of microbiota would be calculated as counts of the pathogen/total counts.
Prevalence of periodontal pathogens (%) in each group_baseline | Baseline
  Four sites will be selected, one per quadrant, based on presence of bleeding during the screening visit. The same sites will be sampled at the follow-up visit. These sites will be isolated with cotton rolls and dried gently with sprayed air. Two consecutive sterile paper points (medium size, Maillefer, Ballaigues, Switzerland) will be inserted as deep as possible into the sulcus, and leave in place for 10 seconds. The paper points will be transferred to a vial containing 1.5 mL of reduced transport fluid (Syed & Loesche, 1972), and pooled with the other paper points.
  The vial will be sent to the laboratory and processed for culture and qPCR. Prevalence would be defined as presence/absence of each pathogen.
Prevalence of periodontal pathogens (%) in each group_6 weeks | 6 weeks
  Four sites will be selected, one per quadrant, based on presence of bleeding during the screening visit. The same sites will be sampled at the follow-up visit. These sites will be isolated with cotton rolls and dried gently with sprayed air. Two consecutive sterile paper points (medium size, Maillefer, Ballaigues, Switzerland) will be inserted as deep as possible into the sulcus, and leave in place for 10 seconds. The paper points will be transferred to a vial containing 1.5 mL of reduced transport fluid (Syed & Loesche, 1972), and pooled with the other paper points.
  The vial will be sent to the laboratory and processed for culture and qPCR. Prevalence would be defined as presence/absence of each pathogen.
Prevalence of periodontal pathogens (%) in each group_12 weeks | 12 weeks
  Four sites will be selected, one per quadrant, based on presence of bleeding during the screening visit. The same sites will be sampled at the follow-up visit. These sites will be isolated with cotton rolls and dried gently with sprayed air. Two consecutive sterile paper points (medium size, Maillefer, Ballaigues, Switzerland) will be inserted as deep as possible into the sulcus, and leave in place for 10 seconds. The paper points will be transferred to a vial containing 1.5 mL of reduced transport fluid (Syed & Loesche, 1972), and pooled with the other paper points.
  The vial will be sent to the laboratory and processed for culture and qPCR. Prevalence would be defined as presence/absence of each pathogen.

CONTACTS AND LOCATIONS:
Overall Officials: David Herrera, Prof, Principal Investigator — University Complutense
Locations (1):
- Faculty of Dentistry, Univesity Complutense, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Data would be made available upon a reasonable request